CLINICAL TRIAL: NCT05781087
Title: Optical Coherence Tomography With Magnetic Resonance Angiography to Assess STEMI Non-culprit Risk
Brief Title: Predicting the Risk of Non-culprit Coronary Artery Disease After a Heart Attack
Acronym: OCT-RISK
Status: Recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other); King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 292740; FS/CRTF/22/24342 (Other Grant/Funding Number: British Heart Foundation)
Record Dates: First submitted 2023-03-09; First posted 2023-03-23 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Coronary Artery Disease; ST Elevation Myocardial Infarction; Ischemic Heart Disease
Keywords: optical coherence tomography; non-culprit; magnetic resonance imaging; cardiac magnetic resonance; STEMI; magnetic resonance angiography; OCT
MeSH Terms: conditions — Coronary Artery Disease; ST Elevation Myocardial Infarction; Myocardial Ischemia | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standard of care: Patients after ST-elevation myocardial infarction with non-culprit coronary artery disease.
  Interventions: Diagnostic Test: Optical coherence tomography and pressure wire assessment; Diagnostic Test: Cardiac magnetic resonance angiogram

INTERVENTIONS:
Diagnostic Test: Optical coherence tomography and pressure wire assessment — Non-culprit coronary arteries
  Other Names: OCT (Abbott); PressureWire X (Abbott)
Diagnostic Test: Cardiac magnetic resonance angiogram — 1.5T
  Other Names: Cardiac MRI

SUMMARY:
Heart attacks caused by the complete blockage of a heart artery are treated by opening it with a stent. However, most people will also have 'non-culprit' narrowings found in their other arteries at this time.

Although in general people do better if these non-culprit narrowings are also treated with stents if they look severe, this process has problems. This is because narrowings that look severe may be stable and not cause any trouble. For these people a stent is a wasted procedure and unnecessary risk. On the other hand, narrowings that are currently left alone because they appear mild, may progress and cause a heart attack.

Participants who have had a heart attack will have a scan from inside the heart arteries during an angiogram (optical coherence tomography, OCT) and a magnetic resonance angiogram (MRA).

If the investigators can show that it is possible to accurately predict which non-culprit narrowings are going to progress and which are going to stabilise, medical professionals may be able to better target their treatments after a heart attack.

ELIGIBILITY:
Inclusion Criteria:

* Successful primary percutaneous coronary intervention (PCI) within the previous week with no major complications at the index procedure
* Bystander disease in a non-culprit vessel planned for clinically indicated staged angiography +/- PCI
* Able to provide written informed consent.

Exclusion Criteria:

* Cardiogenic shock requiring intubation, inotropes or a mechanical support device
* Creatinine clearance <30ml/min
* Prior coronary artery bypass grafting
* Life expectancy less than 3 years
* Pregnancy.
* Target lesion in the left main coronary artery
* Severe calcification or tortuosity that would threaten safe placement of a pressure wire or OCT catheter
* Chronic total occlusion of a major epicardial vessel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after presentation with ST elevation myocardial infarction.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Change in mean fibrous cap thickness measured by optical coherence tomography | 6 months

SECONDARY OUTCOMES:
Change in mean lipid arc measured by optical coherence tomography | 6 months
Presence of thin cap fibroatheroma measured by optical coherence tomography | 6 months
  Plaque with lipid arc >90° and fibrous cap thickness ≤65µm
Change in measures of shear stress made by optical coherence tomography and magnetic resonance angiography | 0 and 6 months
  Comparison between non-invasive and invasively derived measures

OTHER OUTCOMES:
Non-culprit major adverse cardiac events | 6 months and 36 months
  Death, myocardial infarction, ischaemia driven revascularisation
Change in vessel stenosis measured by optical coherence tomography and magnetic resonance angiography | 0, 6 and 36 months
  Comparison between non-invasive and invasively derived measures

CONTACTS AND LOCATIONS:
Overall Officials: Divaka Perera, MD, Principal Investigator — King's College London
Locations (2):
- United Kingdom (2):
  - St Thomas' Hospital, London
  - King's College Hospital, London

IPD SHARING:
Plan to Share IPD: No